CLINICAL TRIAL: NCT03685474
Title: Facing Your Fears in Schools: Implementing a CBT Program for Students With ASD or Other Special Learning Needs
Acronym: FYF-SB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18-0114
Record Dates: First submitted 2018-09-11; First posted 2018-09-26 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Special Learning Needs; Minority Groups
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: In the present study, we will use the measure entitled Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM; Glasgow, 2013) as a framework for planning and implementing FYF-SB in the school environment. The translation of research from controlled research settings to natural environments is often an exceptionally slow process, perhaps because of the emphasis on efficacy. A pragmatic framework such as RE-AIM can hasten the portability of evidenced based intervention to "real-world" practice by focusing on stakeholder feedback and environmental context, in conjunction with intervention development and content.
  We plan to conduct a randomized controlled trial of the FYF-SB intervention across 30 schools within 3 districts. The intervention conditions occur for 1 semester within an academic year. Data will be collected in a pre-post design (before and after the condition of either Facing Your Fears - School Based or Usual Care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facing Your Fears-School Based (FYF-SB) (Experimental): This group will receive the Facing Your Fears - School Based intervention during the fall semester
  Interventions: Behavioral: Facing Your Fears - School Based
- Usual Care (UC) (Active Comparator): This group will receive usual care of anxiety treatment during the fall semester, but will be in the FYF-SB arm the following spring semester.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Facing Your Fears - School Based — Participants receiving FYF-SB will receive cognitive-behavioral treatment (CBT), which is an evidence-based practice (EBP) for treating anxiety in typical youth, within their school setting.
  Other Names: Cognitive Behavioral Treatment
  Arms: Facing Your Fears-School Based (FYF-SB)
Behavioral: Usual Care — Participants receiving usual care will experience no different therapies, strategies, or recommendations other than what would typically be administered within the school setting in the absence of the proposed study.
  Arms: Usual Care (UC)

SUMMARY:
The overall goal of the project is to develop a feasible, effective and sustainable school-based program to manage anxiety in elementary and middle school students with Autism Spectrum Disorder (ASD) and other special learning needs. There are two phases to this Department of Health and Human Services/Health Resources and Services Administration-funded research. In the first phase, there will be engagement of community partners in the process of developing the adapted intervention for implementation in schools. The first phase is ongoing until approximately fall of 2018.

This project is the second phase of this program of research and is focused on piloting and implementing the school-based intervention within 3 local school districts in a systematic and sustainable way - through a "train-the-trainer" model. Primary aims are:

1. to prepare cross-disciplinary teams of School - Based Trainers to conduct three pilot student groups of Facing Your Fears - School Based (FYF-SB) within their own district, with the goal of later training others in their districts to deliver FYF-SB.
2. at the start of the following academic year (2019-2020), within each of the three participating districts, 10 schools will be randomized to one of two conditions for the fall semester: a) FYF-SB or b) Usual Care; and assess implementation and treatment outcomes.

DETAILED DESCRIPTION:
Children with Autism Spectrum Disorder (ASD) are at high risk for developing clinically significant anxiety. Anxiety markedly interferes with peer relationships, family functioning and participation in academic programming. Youth with ASD demonstrate significant reductions in anxiety following participation in treatments rooted in evidence-based practice (EBP) such as cognitive behavior therapy (CBT). The treatment program, Facing Your Fears (FYF), is one such EBP. However, substantial disparities in access to psychiatric services exist, particularly for youth from minority and/or low income families. Schools may be the ideal location to access these services because they represent one of the only consistent resources available to many low resourced families.

The current proposal is innovative for several reasons: (1) There are very few published studies examining the effectiveness of treatments for children with ASD and anxiety in schools, and none that have focused on under-resourced communities; (2) There are no known studies that have identified students for an intervention program according to special education eligibility criteria, combined with other inclusion criteria, an approach which will likely serve more students, and in turn, potentially increase the feasibility of FYF-SB; (3) a "train the trainer" model will result in increased capacity for low resourced schools to serve underserved youth; and (4) Finally, the current study is one of the first to examine organizational constructs that are potentially associated with adoption of FYF-SB, the results of which would help determine critical next steps in implementation research.

Overview of Facing Your Fears (FYF): The clinical version of FYF is a 14-week, family-focused CBT group intervention (1 ½ hours each session) aimed toward managing anxiety in children ages 8-14 with high-functioning ASD. FYF is composed of three books (e.g., facilitators, parents and children) and a digital versatile disc (DVD). The 14 weeks are divided into two, seven-session intervention blocks: (1) an introduction to anxiety symptoms with an emphasis on the individual expression of anxiety symptoms, as well as an introduction to common CBT strategies, and (2) a focus on using specific tools and strategies (i.e. deep breathing, positive coping statements and graded exposure--facing fears a little at a time) to improve emotion regulation and manage anxiety symptoms. Although FYF was originally developed for youth with ASD, there is no mention of ASD in the curriculum, as the focus is exclusively on management of anxiety. Importantly, careful attention was paid to the delivery of core concepts, given the social, communicative and cognitive challenges of youth with ASD (Moree & Davis, 2010). The use of written worksheets, multiple choice lists, emphasis on creative and varied outlets for expression, use of video modeling and a focus on strengths and talents make FYF ideal for students with special learning needs.

Facing Your Fears: School-Based (FYF-SB): FYF-SB will be very similar to FYF, but will be modified for delivery in school settings. Phase 1 study, currently in completion, will enable input to be obtained from school personnel, district leaders and parents as a way to determine the best ways to adapt the intervention for schools. Thus the logistical details of how the intervention will be offered to students within each participating school district has been discussed in detail with each of the 3 participating districts' leaders and key personnel.

Research Methods:

Aim 1: Implement FYF-SB in school settings and assess effectiveness Train teams of School-Based Trainers to deliver FYF-SB to students and then train other professionals. Cross-disciplinary school providers will be selected by district administrators to serve as School-Based Trainers ("Trainers"). The Trainers (10 per district will be recruited to account for attrition) will be trained to deliver FYF-SB to small groups of 2-4 students with ASD or special learning needs and anxiety during the initial pilot study of the intervention. These school-based professionals will become the "trainers" for their own individual districts, once they have completed their own training activities.

Becoming a School-Based Trainer for the project will involve: (1) Attending a two day interactive workshop, focused on the principles of CBT and core components of FYF-SB. The training will take place during non-academic periods. The workshop will be interactive and dynamic (per Becker & Stirman, 2011), including group discussion, experiential exercises, small group activities and videotaped examples. (2) Participating in ongoing consultation and technical assistance throughout at least one academic year with the research team; (3) Meeting expectations for fidelity on the intervention (average fidelity score >80%, based on a minimum of 3 observations). School-Based Trainers who do not meet the fidelity requirements will be asked to participate in additional training in order to continue in that role. School-Based Trainers can always decide to become School-Based Providers (delivering the intervention to students, but not train others) instead and/or can always decide to participate in the project or not, as their participation is purely voluntary.

Aim 2 - Randomize schools across three districts to either FYF-SB or Usual Care (UC) and assess outcomes. The second part of the implementation phase is to evaluate the effectiveness of FY-SB; thus, a small randomized controlled trial will be conducted across school districts. Trainers will participate in "train the trainer" activities to prepare them for training their own school teams in the delivery of FYF-SB. Ten schools across each district will be randomized to either FYF-SB or Usual Care. The five schools (and their School-Based Trainers and School Providers) that are randomized to FYF-SB, will receive training and consultation from the Trainers, and school providers will deliver FYF-SB to a cohort of target students. Schools that are randomized to Usual Care will identify students who meet inclusion criteria for the study, and will take pre- and post-wait assessment data. The UC Sites will have the opportunity to deliver FYF-SB the next semester if they so choose. Investigators anticipate 60 providers will be trained across the districts.

FYF-SB will be delivered in elementary and middle schools across three main districts: Cherry Creek School District (CCSD), Denver Public Schools (DPS) and Littleton Public Schools (LPS). All three districts have economically and ethnically diverse student bodies. DPS is the largest district of the three, with 93 elementary schools. The student population in DPS is more than 56% Hispanic and 14% African American. CCSD has 42 elementary schools and LPS has 13 elementary schools; all three districts also have racially and ethnically diverse schools, as well as low-income populations. All of the districts have large populations of students with ASD. The districts have all expressed strong interest in this project, and have been actively involved in Phase 1.

The results of this study will provide information about the feasibility and acceptability of implementing a school-based cognitive behavioral intervention aimed at reducing the impact of anxiety on school functioning for students with ASD. If this method of treatment delivery proves to be feasible and potentially effective, it has the potential to improve access to mental health support for youth who do not have ready access to specialists in the medical community and for whom mental health supports are provided primarily in educational settings.

Successful completion of this study will result in a sustainable school based treatment program to manage anxiety in students with ASD or other special learning needs. Successful implementation and treatment outcomes will result in improved internal capacity of schools to treat the significant and interfering anxious symptoms of underserved students with ASD or other special learning needs. Reductions in interfering anxiety symptoms for high risk, underserved students with ASD or other special learning needs, can lead to marked improvements in school functioning. The results of this study will also help to identify factors that may influence the implementation of FYF-SB (e.g., organizational constructs, principal leadership), which may help determine critical next steps in implementation research in school settings.

ELIGIBILITY:
Inclusion Criteria:

1. Estimated Verbal intelligence quotient (IQ) of 80 or above as determined by the Weschler Abbreviated Scales of Intelligence (WASI), or an equivalent measure administered within the past three years; or presents with achievement scores in school records that suggest average-low average-borderline intellectual functioning
2. Clinically significant anxiety symptoms as defined by significant elevations on either the SCARED, or PRAS-ASD, according to either student, parent, or teacher report
3. Currently staffed into special education with an individualized education plan (IEP) or 504 with one of the following eligibility categories: autism, other health impairment, emotional disturbance, specific learning disabilities, multiple disabilities or other speech/language impairment; OR currently identified as at risk and in need of Response to Intervention (RTI) consultation and not yet found to be eligible for special education services OR currently in the process of completing the educational eligibility evaluation
4. Significant deficits in reciprocal social behavior as defined by a Total T Score on the Social Responsive Scale Version 2 (SRS-2) of 60 or above
5. Lives with parent/guardian who can provide consent for participation.

Exclusion Criteria:

(1) Presentation of psychosis, severe aggressive behavior, or other severe clinical symptoms that require more intensive treatment such as day treatment or hospitalization

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 389 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Reduction in symptoms of anxiety of the participant as measured by scores from the teacher - completed questionnaire, The School Anxiety Scale (SAS). | 13 weeks
  The School Anxiety Scale (Lyneham et al. 2008) is a 16 item teacher-reported measure of anxiety designed to assess the behavior of children at school from 5 to 12 years of age. Items are answered on a four-point scale. This measure provides a total score for anxiety, with scores ranging from 0 - 48. Two subscales are also calculated, reflecting social anxiety and generalized anxiety.
  This measure will be completed by teachers before and after study treatment.
Reduction in symptoms of anxiety of participants as measured by scores from the parent-completed questionnaire, Parent-Rated Anxiety Scale for ASD (PRAS-ASD). | 13 weeks
  The Parent - Rated Anxiety Scale for ASD (Scahill et al.) is a 25 item, parent report measure created to assess anxiety in youth with ASD. This measure has good test - retest reliability of 0.88 and 0.86, and strong convergent validity with other anxiety measures (0.83).
  This measure will be completed by parents before and after study treatment.
Reduction in symptoms of anxiety of participant as measured by scores from parent -, and self - completed questionnaire, Screening for Childhood Anxiety and Related Emotional Disorders (SCARED). | 13 weeks
  Screening for Childhood Anxiety and Related Emotional Disorders (Birmaher et al, 1999) if a 40 - item inventory of statements that assess five types of anxiety experienced by children and adolescents, to be completed separately by parents and students. A total score, as well as cutoffs for specific domains on anxiety (e.g., social, generalized) are obtained. A total score of 25 or higher is considered to be clinically significant. Youth who obtain a score above the clinical cutoff for the total score or for 1 or more domains are eligible.
  This measure will be completed by parents and students before and after study treatment.
Reduction in symptoms of anxiety of participants as measured by scores from parent - completed questionnaire, The Social Responsiveness Scale, Second Edition (SRS-2). | 13 weeks
  The Social Responsiveness Scale (Constantino & Gruber, 2012) is a parent - reported 65 - item questionnaire that uses a 4 - point Likert scale to assess behaviors associated with ASD. It included five subscales: awareness, cognition, communication, motivation, and autistic mannerisms. Higher scores suggest greater impairment. The SRS is commonly used in autism research, has good reliability, and is valid across cultures (Bolte et al., 2008).
  This measure will be completed by parents before and after study treatment.
Reduction in symptoms of anxiety of participants as measured by scores from parent -, and teacher - completed questionnaire, Emotion Regulation Checklist (ERC). | 13 weeks
  The Emotion Regulation Checklist (Shields & Cicchetti, 1997) is a 24 - item parent/teacher report measure that provides information regarding a child's typical responses to emotionally intense experiences. The instrument has good reliability and validity across adult informants and provides indices regarding the child's ability to modulate and express affect in a manner that is context - appropriate. The ERC has been shown to be sensitive to change in effectiveness studies of CBT protocols with anxious youth (Suveg, Kendall, Comer, & Robin, 2006).
  This measure will be completed by teachers and parents before and after study treatment.
Classroom attendance | 13 weeks
  Teachers will track participants' daily attendance, including late arrivals and amount of time spent outside of classroom. Progression will be tracked for any trends before, during, and after study participation.

SECONDARY OUTCOMES:
Protocol adherence as measured by fidelity checklist. | 13 weeks
  The Treatment fidelity/acceptability checklist will be used to assess facilitators' adherence to protocol. The measure is a checklist that assesses the presence / absence of core treatment components on a session - by - session basis, while simultaneously assessing usefulness and acceptability. Because school providers, students, and parents will complete this measure, we will be able to cross - check adherence and utility of core activities.
Emotion Dysregulation Inventory Scores: Dysphoria | Baseline, 13 Weeks
  The Emotion Dysregulation Inventory dysphoria subscale measures emotional dysregulation and dysphoria. Possible scores range from 6 to 30, with higher scores indicating a worse outcome. This outcome measure was added via a protocol amendment in July 2019.
Emotion Dysregulation Inventory Scores: Reactivity | Baseline, 13 Weeks
  The Emotion Dysregulation Inventory reactivity subscale measures emotional dysregulation and reactivity. Possible scores range from 7 to 35, with higher scores indicating a worse outcome. This outcome measure was added via a protocol amendment in July 2019.
Teacher Concern Inventory: Time Management Subscale | Baseline, 13 Weeks
  The Teacher Concern Inventory measures educator stress and concern. 5 subscales are used: Time Management, Work Stressors, Professional Distress, Discipline and Motivation, and Professional Investment. The possible scores for the Time Management subscale range from 8 to 40, with higher scores indicating a worse outcome. This outcome measure was added via a protocol amendment in July 2019.
Teacher Concern Inventory: Work Stressors | Baseline, 13 Weeks
  The Teacher Concern Inventory measures educator stress and concern. 5 subscales are used: Time Management, Work Stressors, Professional Distress, Discipline and Motivation, and Professional Investment. The possible scores for the Work Stressors subscale range from 6 to 30, with higher scores indicating a worse outcome. This outcome measure was added via a protocol amendment in July 2019.
Teacher Concern Inventory: Professional Distress | Baseline, 13 Weeks
  The Teacher Concern Inventory measures educator stress and concern. 5 subscales are used: Time Management, Work Stressors, Professional Distress, Discipline and Motivation, and Professional Investment. The possible scores for the Professional Distress subscale range from 5 to 25, with higher scores indicating a worse outcome. This outcome measure was added via a protocol amendment in July 2019.
Teacher Concern Inventory: Discipline and Motivation | Baseline, 13 Weeks
  The Teacher Concern Inventory measures educator stress and concern. 5 subscales are used: Time Management, Work Stressors, Professional Distress, Discipline and Motivation, and Professional Investment. The possible scores for the Discipline and Motivation subscale range from 6 to 30, with higher scores indicating a worse outcome. This outcome measure was added via a protocol amendment in July 2019.
Teacher Concern Inventory: Professional Investment | Baseline, 13 Weeks
  The Teacher Concern Inventory measures educator stress and concern. 5 subscales are used: Time Management, Work Stressors, Professional Distress, Discipline and Motivation, and Professional Investment. The possible scores for the Professional Investment subscale range from 4 to 20, with higher scores indicating a worse outcome. This outcome measure was added via a protocol amendment in July 2019.

OTHER OUTCOMES:
Exploratory measure to assess plans for long-term maintenance of the program. | 13 weeks
  The Evidence - Based Practice Attitude Scale (EBPAS; Aarons et al., 2004) is a 15 - item scale measured on a five point scale that assesses general attitude towards the adoption of EBP. There are four subscales that measure appeal, requirements, openness, and divergence. Subscale and total scores can be calculated. The EBPAS has demonstrated strong internal consistency. This measure will be used in order to plan for long-term maintenance and sustainability of the program.
Exploratory measure to assess individual schools' organizational and training climates through the Organizational Readiness for Change (ORC) measure. | 13 weeks
  The ORC (Lehman, et al. 2002) is a 129 item scale that measures organizational characteristics on a five point Likert scale, across five domains: motivation, resources, staff attributes, organizational climate, and training climate. This measure will be used to assess the potential for program sustainability within each participating school.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Reaven, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reaven J, Cosgrove KT, Losh A, Nickles S, Kerns CM, Pickard K, Blakeley-Smith A, Hayutin L, Meyer AT, Middleton C, Reyes NM, Boles RE. Facing your fears in schools: using the ADIS/ASA to characterize anxiety and intervention outcomes in students with autism or suspected autism. Front Psychiatry. 2025 Jul 23;16:1569435. doi: 10.3389/fpsyt.2025.1569435. eCollection 2025. PMID 40778329

DOCUMENTS (1):
  • Informed Consent Form (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03685474/ICF_000.pdf